CLINICAL TRIAL: NCT03657810
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study to Determine the Efficacy and Safety of CL-108 5 mg (Hydrocodone 5 mg/Acetaminophen 325 mg/Promethazine 12.5 mg) as a Treatment for Moderate-to-Severe Acute Pain and the Prevention of Opioid-Induced Nausea and Vomiting (OINV) Following Orthopedic Surgery
Brief Title: A Controlled Study to Determine the Efficacy and Safety of CL-108 5 mg for Acute Pain and the Prevention of OINV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charleston Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCT-018
Record Dates: First submitted 2017-12-05; First posted 2018-09-05 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Pain; Nausea; Vomiting
Keywords: Pain; Nausea; Vomiting
MeSH Terms: conditions — Pain; Nausea; Vomiting | interventions — Hydrocodone; Acetaminophen; Promethazine; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CL-108 5 mg (Experimental): Hydrocodone 5 mg/APAP 325 mg/promethazine 12.5 mg (CL-108 5 mg) bi-layered tablet
  Interventions: Drug: CL-108 5 mg
- Norco (Active Comparator): hydrocodone 5 mg/APAP 325 mg
  Interventions: Drug: Norco
- Placebo (Placebo Comparator): Placebo 0 mg matching CL-108
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CL-108 5 mg — hydrocodone 5 mg/APAP 325 mg/promethazine 12.5 mg
  Other Names: hydrocodone bitartrate/ acetaminophen/ promethazine hydrochloride
  Arms: CL-108 5 mg
Drug: Norco — hydrocodone 5 mg/APAP 325 mg
  Other Names: hydrocodone bitartrate/ acetaminophen
  Arms: Norco
Drug: Placebo — Placebo matching CL-108
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
To determine the analgesic efficacy of CL-108 5 mg by comparison with placebo and the anti-emetic efficacy of CL-108 5 mg by comparison with hydrocodone 5 mg/acetaminophen 325 mg.

DETAILED DESCRIPTION:
Adult patients with moderate or severe pain after bunionectomy will be randomized to CL-108 5 mg (hydrocodone 5 mg/acetaminophen 325 mg/ promethazine 12.5 mg), hydrocodone 5 mg/ acetaminophen 325 mg, or placebo under double-blind conditions. Over 48 hours they will use the assigned study medication and assess pain intensity, nausea, and vomiting. Uses of supplementary analgesic and antiemetic medications will be documented. Patient responses and adverse effects will also be documented during the 5-day outpatient period, too.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Signed informed consent form obtained at screening prior to any procedures being performed.
* Gender: Male or non-pregnant and non-lactating female.
* Age: 18 years or older at time of consent.
* Foot condition: Primary unilateral first metatarsal bunionectomy (osteotomy and internal fixation) with no additional collateral procedures.
* Pain Severity: Presence of moderate or severe pain on a categorical pain intensity scale at Baseline
* Pain Confirmation: On the 0-10 numerical pain intensity scale at Baseline.
* Diary Completion: Be willing and able to record safety and efficacy ratings in the Diaries.
* Safe Transportation Home: Patient must have arrangements for transportation home from the research center accompanied by a responsible adult.

Exclusion Criteria:

* Medical condition: Presence of a serious medical condition, intolerance to NSAIDs, or any other medical condition which, in the opinion of the Investigator, makes the patient unsuitable for participation.
* Infection: Acute infection of the surgical site at the time of surgery that could confound post-surgical evaluation.
* Drug Allergy: History of hypersensitivity to an opioid drug (such as hydrocodone), promethazine, acetaminophen, NSAID (such as ibuprofen or aspirin), midazolam, propofol, mepivacaine, ropivacaine or ketorolac.
* Confounding and Contraindicated Drugs: Other than protocol-permitted medications administered pre-operatively or during surgery: use within 14 days before or during the surgical procedure of any systemic corticosteroid or use within 24 hours or during the surgical procedure of any confounding prescription or non-prescription drug or any drug contraindicated with hydrocodone, acetaminophen, or promethazine. [Note: Antibiotic for endocarditis prophylaxis (except if known to cause nausea) and aspirin (ASA) ≤ 325 mg for cardiovascular prophylaxis are permitted during the study.] History of consuming more than 2 alcoholic drinks per day every day for the last month or a positive urine test for opiates, benzodiazepines, barbiturates, tetrahydrocannabinol, methamphetamines, cocaine, oxycodone, cotinine at screening or the morning of surgery will exclude the patient from the trial.
* Investigational Drug Use: Use of an investigational drug within the past 30 days.
* Participated in Study: Previous participation in this study.
* Pregnancy, Lactation: Women who are pregnant or lactating.
* Compliance: Inability to swallow capsules whole.
* Participant relationship: Employee at the research center, employee of the Principal Investigator, Sub-Investigators, or sponsor or relative of the Investigator, Sub-Investigators or research staff who is involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Schachtel, MD, Study Director — Charleston Laboratories, Inc
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - Chesapeake, Pasadena, Maryland
  - Optimal Research, Austin, Texas
  - Endeavor Clinical Research, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Charleston Website — http://www.charlestonlabs.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, double-blind, randomized, placebo- and active-controlled, multiple-dose study conducted at different research centers in the United States
Pre-assignment Details: A total of 349 subjects were enrolled into the study, 128 were Screen Failed and 221 were Randomized, 209 were Completed the study and 12 subjects were discontinued.
Groups:
- CL-108: Hydrocodone 5 mg/acetaminophen (APAP) 325 mg/promethazine 12.5 mg (CL-108 5 mg) bi-layered tablet
  CL-108 5 mg: hydrocodone 5 mg/APAP 325 mg/promethazine 12.5 mg
Period: Overall Study
Arm/Group | CL-108 | Norco | Placebo
Started | 87 | 90 | 44
Completed | 82 | 86 | 41
Not Completed | 5 | 4 | 3
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lack of Efficacy | 4 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Not provided | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized patients who received at least 1 dose of study medication constituted the Safety Population.
Groups:
- CL-108: Hydrocodone 5 mg/APAP 325 mg/promethazine 12.5 mg (CL-108 5 mg) bi-layered tablet
  CL-108 5 mg: hydrocodone 5 mg/APAP 325 mg/promethazine 12.5 mg
- Total: Total of all reporting groups
Arm/Group | CL-108 | Norco | Placebo | Total
Number analyzed (Participants) | 87 | 90 | 44 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.97) | 43.5 (14.74) | 47.2 (13.40) | 44.2 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 77 | 40 | 192
  Male | 12 | 13 | 4 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 22 | 9 | 58
  Not Hispanic or Latino | 60 | 68 | 35 | 163
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 12 | 12 | 8 | 32
  White | 69 | 73 | 33 | 175
  More than one race | 2 | 2 | 0 | 4
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 87 | 90 | 44 | 221
Weight [Mean (Standard Deviation); unit: kg] | 79.19 (23.427) | 74.56 (18.054) | 81.86 (18.827) | 77.83 (20.592)
Height [Mean (Standard Deviation); unit: cm] | 164.94 (9.457) | 165.09 (9.133) | 164.45 (8.256) | 164.90 (9.060)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.88 (6.876) | 27.29 (5.549) | 30.26 (6.358) | 28.51 (6.333)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With OINV Over 48 Hours
Description: Number and Percentage of participants With opioid-induced nausea and vomiting (OINV) who experienced any Vomiting / use of Anti-Emetic Medication Over 48 Hours
Time Frame: Up to 48 hours
Population: Intent-to-Treat (ITT) Population: The ITT Population comprised all patients who were randomized and who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
Participants | 8 | 31 | 4
Statistical Analysis 1: Comparison: CL-108 vs Norco; Test type: Superiority; p < 0.001, Regression, Logistic — Type III P-Value are from the likelihood ration test from the logistic regression model with factors of treatment, gender, and investigator

2. Primary Outcome: The Sum of Pain Intensity Differences (on PI-NRS) Over 48 Hours (SPID48)
Description: The SPID48 endpoint is calculated from the PI-NRS values at baseline, every 30 minutes until hour 12, then every hour (when awake) until hour 48 as follows:
  * Each subsequent PI-NRS value is subtracted from the baseline PI-NRS value.
  * Each difference is weighted by the elapsed time from the previous PI-NRS value to the current one.
  * The weighed differences are summed to yield the SPID48.
  Summed pain intensity differences over 48 hours (SPID48) will be compared for patients treated with CL-108 5 mg and those treated with placebo. Pain intensity will be measured on a 0-10 Pain Intensity Numerical Rating Scale (PI-NRS), where 0 is "no pain" and 10 is "severe pain".
Time Frame: Up to 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
score on a scale | 108.5 (80.66) | 94.8 (69.53) | 78.7 (62.66)
Statistical Analysis 1: Comparison: CL-108 vs Norco; Test type: Superiority; p = 0.052, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Patients With Complete Absence of OINV (no Nausea, no Vomiting, and no Use of Anti-emetic Medication) Over 48 Hours
Description: Percentage of patients with complete absence of OINV (no nausea, no vomiting, and no use of anti-emetic medication) over 48 hours comparing CL-108 5 mg to hydrocodone 5 mg/APAP 325 mg)
Time Frame: Up to 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
Participants | 50 | 34 | 27

4. Secondary Outcome: Percentage of Patients With Any Vomiting Over 48 Hours
Description: Percentage of patients with any vomiting over 48 hours, comparing CL-108 5 mg to hydrocodone 5 mg/APAP 325 mg
Time Frame: Up to 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
Participants | 3 | 19 | 2

5. Secondary Outcome: Percentage of Patients With Any Nausea Over 48 Hours
Description: Percentage of patients with any nausea over 48 hours, comparing CL-108 5 mg to hydrocodone 5 mg/APAP 325 mg
Time Frame: Up to 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
Participants | 36 | 55 | 15

6. Secondary Outcome: Percentage of Patients With Any Nausea or Vomiting Over 48 Hours
Description: Percentage of patients with any nausea or vomiting over 48 hours, comparing CL-108 5 mg to hydrocodone 5 mg/APAP 325 mg
Time Frame: Up to 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
Participants | 37 | 55 | 16

7. Secondary Outcome: Percentage of Patients With Any Post-discharge Nausea and Vomiting (PDNV)
Description: Percentage of patients with any Post-discharge Nausea and Vomiting (PDNV) over Days 3 to 7
Time Frame: Day 3 to 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
Participants | 9 | 12 | 6

8. Secondary Outcome: Number of Doses of Study Medication Taken Over Days 3to7
Description: Number of doses of study medication taken over Days 3 to 7
Time Frame: Day3 to Day7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
doses | 10.0 (7.05) | 8.4 (7.30) | 6.2 (5.70)

9. Secondary Outcome: Number of Doses of Study Medication Taken Per Day Over Days 3to7
Description: Number of doses of study medication taken per day over Days 3 to 7
Time Frame: Day3 to Day7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: doses per day
Arm/Group | CL-108 | Norco | Placebo
Number analyzed (Participants) | 87 | 90 | 44
doses per day
  Number of Doses of Study Medication Taken over Day 3 | 3.0 (1.60) | 2.4 (1.83) | 2.1 (1.59)
  Number of Doses of Study Medication Taken over Day 4 | 2.1 (1.65) | 1.9 (1.70) | 1.4 (1.45)
  Number of Doses of Study Medication Taken over Day 5 | 1.9 (1.81) | 1.7 (1.73) | 1.1 (1.40)
  Number of Doses of Study Medication Taken over Day 6 | 1.8 (1.77) | 1.5 (1.72) | 1.0 (1.16)
  Number of Doses of Study Medication Taken over Day 7 | 1.1 (1.46) | 0.9 (1.29) | 0.6 (1.06)

ADVERSE EVENTS:
Time Frame: Up to Visit 3 (Approximately 8 days after surgery)
Description: A drug-related (TEAE) Treatment-emergent adverse event is defined as a TEAE with a relatedness of Possible or Probable. A subject is counted once in the most severe category if the subject reported one or more events, but different severity.
Arm/Group | CL-108 | Norco | Placebo
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/90 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/87 | 0/90 | 0/44
Other Adverse Events (participants affected / at risk) | 80/87 | 79/90 | 37/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CL-108 (N=87) | Norco (N=90) | Placebo (N=44)
DEEP VEIN THROMBOSIS RIGHT CALF (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CL-108 (N=87) | Norco (N=90) | Placebo (N=44)
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 38 | 54 | 17
Dry mouth (Gastrointestinal disorders) | 31 | 16 | 8
Constipation (Gastrointestinal disorders) | 23 | 24 | 4
Vomiting (Gastrointestinal disorders) | 3 | 20 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 3
Asthenia (General disorders) | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 2
Infusion site extravasation (General disorders) | 0 | 2 | 0
Administration site nodule (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 46 | 40 | 9
Headache (Nervous system disorders) | 22 | 26 | 12
Dizziness (Nervous system disorders) | 22 | 23 | 6
Disturbance in attention (Nervous system disorders) | 10 | 7 | 3
Syncope (Nervous system disorders) | 2 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 7 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 1
Polyuria (Renal and urinary disorders) | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 21 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03657810/Prot_SAP_000.pdf